CLINICAL TRIAL: NCT06104670
Title: The Effect of Synaquell™ on Objective Measures of Brain Health in Male and Female Youth Contact Sport Athletes
Brief Title: The Effect of Synaquell™ in Contact Sport Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Sanford Health (Other)
Responsible Party: Principal Investigator, Mario Hevesi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-005242
Record Dates: First submitted 2023-10-20; First posted 2023-10-27 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Ice Hockey; Cognitive Function; Cognition Brain Supplement; Contact Sport Athletes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study staff responsible for distributing SynaquellTM will not be blinded to the intervention, but all subjects and other study staff will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental: Synaquell Male Group (Experimental): Male youth hockey players will receive the dietary supplement Synaquell, twice-daily during the hockey season. Due to difference in game rules and playing styles, males and females will be treated as two separate arms of the research protocol.
  Interventions: Dietary Supplement: Synaquell(TM)
- Placebo Comparator: Placebo Male Group (Placebo Comparator): Male youth hockey players will receive the placebo twice-daily, during the hockey season. Due to difference in game rules and playing styles, males and females will be treated as two separate arms of the research protocol.
  Interventions: Dietary Supplement: Placebo
- Experimental: Synaquell Female Group (Experimental): Female youth hockey players will receive the dietary supplement Synaquell, twice-daily during the hockey season. Due to difference in game rules and playing styles, males and females will be treated as two separate arms of the research protocol.
  Interventions: Dietary Supplement: Synaquell(TM)
- Placebo Comparator: Placebo Female Group (Placebo Comparator): Female youth hockey players will receive the placebo twice-daily, during the hockey season. Due to difference in game rules and playing styles, males and females will be treated as two separate arms of the research protocol.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synaquell(TM) — 7.9 grams (1 scoop) of Synaquell powder mixed with 12 ounces of water two times per day for the duration of the sport season. The daily amount taken by each participant is (15.8 grams).
  Arms: Experimental: Synaquell Female Group; Experimental: Synaquell Male Group
Dietary Supplement: Placebo — 7.9 grams (1 scoop) of placebo powder mixed with 12 ounces of water two times per day for the duration of the sport season. The daily amount taken by each participant is (15.8 grams). The placebo looks, smells, and tastes like Synaquell but does not contain active ingredient.
  Arms: Placebo Comparator: Placebo Female Group; Placebo Comparator: Placebo Male Group

SUMMARY:
This research is being done to investigate the dietary supplement, Synaquell (TM), for effects on brain function in youth contact sport athletes.

DETAILED DESCRIPTION:
This randomized clinical trial will compare a brain health supplement (Synaquell) with placebo in both male and female ice hockey players over the course of an entire season. The repeated measure design will compare pre- and post-season objective brain health parameters, including quantitated EEG (Neurocatch), blood & saliva biomarkers, impact monitoring mouthguard, and a rapid number naming test (King Devick).

ELIGIBILITY:
Inclusion Criteria:

* Fluent English Speakers
* Medically cleared to play contact sport

Exclusion Criteria:

* An allergy to the ingredients of Synaquell™ or the placebo (ingredients listed on page
* Clinically documented hearing issues,
* In-ear hearing aid or cochlear implant
* Implanted pacemaker or defibrillator
* Metal or plastic implants in skull
* Lack of verbal fluency in the English language
* History of seizures
* Allergy to rubbing alcohol or EEG gel
* Pregnancy

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in N100 Amplitude | Baseline, Postseason (approximately 6 months).
  Obtained by EEG recording of N100 potential amplitude. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores. Changes in brain vital sign scores are depicted within a radar plot format, with the transformation process preserving the essential ERP results but enabling practical, simplified interpretation.
Change in N100 Latency | Baseline, Postseason (approximately 6 months).
  Obtained by EEG recording of N100 potential latency. Increased latencies are indicative of slower responses. Obtained by EEG recording of N100 potential amplitude. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores. Changes in brain vital sign scores are depicted within a radar plot format, with the transformation process preserving the essential ERP results but enabling practical, simplified interpretation.
Change in P300 Amplitude | Baseline, Postseason (approximately 6 months).
  Obtained by EEG recording of P300 potential amplitude. Increased amplitudes are indicative of larger signals. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores. Changes in brain vital sign scores are depicted within a radar plot format, with the transformation process preserving the essential ERP results but enabling practical, simplified interpretation.
Change in P300 Latency | Baseline, Postseason (approximately 6 months).
  Obtained by EEG recording of P300 potential latency. Increased latencies are indicative of slower responses. This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores. Changes in brain vital sign scores are depicted within a radar plot format, with the transformation process preserving the essential ERP results but enabling practical, simplified interpretation.
Change in N400 Amplitude | Baseline, Postseason (approximately 6 months).
  Obtained by EEG recording of N400 potential amplitude. Increased amplitudes are indicative of larger signals.This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores. Changes in brain vital sign scores are depicted within a radar plot format, with the transformation process preserving the essential ERP results but enabling practical, simplified interpretation.
Change in N400 Latency | Baseline, Postseason (approximately 6 months).
  Obtained by EEG recording of N400 potential latency. Increased latencies are indicative of slower responses.This measures is subsequently linearly transformed to a standardized score on a 0-100 scale, with larger peak amplitudes and shorter peak latencies resulting in higher scores. Changes in brain vital sign scores are depicted within a radar plot format, with the transformation process preserving the essential ERP results but enabling practical, simplified interpretation.
Change in blood biomarker: NfL | Baseline, postseason (approximately 6 months).
  Blood will be at a biomarker level. We will investigate the biomarker neurofilament light (NfL). BDNF. The biomarker will be measured in Nanograms per Milliliter (ng/ml).
Change in blood biomarker SNCB. | Baseline, postseason (approximately 6 months).
  Blood will be at a biomarker level and B-Synuclein will be investigated. The biomarker will be measured in Nanograms per Milliliter (ng/ml).
Change in blood biomarker vWF. | Baseline, postseason (approximately 6 months).
  Blood will be at a biomarker level and Von Willebrand Factor (vWF) will be investigated. The biomarker will be measured in Nanograms per Milliliter (ng/ml).
Change in blood biomarker SNCA. | Baseline, postseason (approximately 6 months).
  Blood will be at a biomarker level and A-Synuclein (SNCA) will be investigated. The biomarker will be measured in Nanograms per Milliliter (ng/ml).
Change in blood biomarker BDNF. | Baseline, postseason (approximately 6 months).
  Blood will be at a biomarker level and Brain Derived Neurotrophic Factor (BDNF) will be investigated. The biomarker will be measured in Nanograms per Milliliter (ng/ml).

SECONDARY OUTCOMES:
Change in King-Devick Test (KDT) scored | Baseline, postseason (approximately 6 months).
  A rapid number-naming test that requires individuals to read 3 numbered patters aloud as fast as possible, the resulting time if the KDT score. The post-season score is compared to the pre-season baseline. An increase in the number of seconds required to read the 3 number patterns is considered to be significant.
Impact Monitor Mouthguard Acceleration | Beginning of practice to last game (approximately 6 months).
  The Impact monitor mouthguard measures head acceleration.
Impact Monitor Mouthguard Rotation | Beginning of practice to last game (approximately 6 months).
  The Impact monitor mouthguard measures rotation of the head.
Impact Monitor Mouthguard Head Impacts | Beginning of practice to last game (approximately 6 months).
  The Impact monitor mouthguard measures the number of head impacts.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Hevesi, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No